CLINICAL TRIAL: NCT03517098
Title: Enhanced Recovery After Surgery (ERAS) Pathway for Primary Hip and Knee Arthroplasty: a Prospective, Controlled, Randomized Clinical Trial
Brief Title: Enhanced Recovery After Surgery (ERAS) Pathway for Primary Hip and Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Associate professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERAS180424
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Arthroplasty, Replacement, Hip, Knee
Keywords: Enhanced recovery after surgery; General anesthesia; Total hip arthroplasty; Total knee arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ERAS group (Experimental): Patients will be treated with the ERAS pathway
  Interventions: Procedure: The ERAS group
- The non-ERAS group (Other): Patients undergoing THA or TKA will receive conventional care.
  Interventions: Procedure: The non-ERAS group

INTERVENTIONS:
Procedure: The ERAS group — ERAS pathway for orthopedic surgeons:
  1. Shortened preoperative fasting from intake.
  2. Preoperative tranexamic acid administration.
  3. No indwelling catheters.
  4. No tourniquet used for TKA.
  5. No drainage tube.
  6. Application of the low molecular heparin 6 hours after the operation.
  ERAS pathway for anesthesiologist:
  1. Intravenous 20 mg of dexamethasone before anesthetic induction.
  2. Anesthesia will be induced with small dose of long-acting opioids such as sulfentanil, or without long-acting opioids at all.
  3. Laryngeal mask for airway.
  4. Anesthesia will be maintained with short-acting anesthetic agents such as desflurane, sevoflurane, or propofol, with continuous remifentanil , and BIS value will be kept between 40 to 60 during procedure.
  5. Incision infiltration with 40-50ml of 0.2% ropivacaine, and no patient controlled intravenous analgesia devices will be applied.
  Arms: The ERAS group
Procedure: The non-ERAS group — Patients undergoing THA or TKA will receive conventional care according to different participating center, and there's no standard protocol for pre-operative management, anesthetic technique or medication choice, postoperative analgesia or food intake, or catheters indwelling.
  Arms: The non-ERAS group

SUMMARY:
As the world goes into the aging society, the number of total hip and total knee arthroplasty (THA and TKA) will increase fast. It's important to develop strategies to improve the quality of healthcare and get earlier recovery and better outcome for patients undergoing THA and TKA. Enhanced recovery after surgery (ERAS) pathways have been reported to promote faster recovery in some clinical settings, but most of them are retrospective cohort study. We hypothesized that ERAS pathway could provide better recovery than current routine clinical practice for patients undergoing primary THA or TKA.

This trial is a prospective, open-labelled, randomized controlled trial that will test, for length of stay (LOS) in hospital, the superiority of ERAS pathway as compared with current clinical practice. A total of 604 patients undergoing primary THA or TKA will be randomized to allocate either ERAS pathway (ERAS group) or conventional care according to different participating center (non-ERAS group). The primary outcome is LOS in hospital. Secondary outcomes include Postoperative LOS, all-cause mortality by 30 days after operation, in-hospital complications, mobilization, postoperative pain evaluation, total in-hospital cost, and readmission rate by 30 days after discharge from the hospital.

DETAILED DESCRIPTION:
Total joint arthroplasty is a definitive treatment for end-stage osteoarthritis of the hip and knee, which is increased as the world goes into the aging society. It was reported that 0.33 million total hip arthroplasty (THA) and 0.7 million total knee arthroplasty (TKA) were performed in the United States annually, and the demand for the procedures were estimated to 0.57 million and 3.48 million per year in 2030, respectively. It's important to find strategies to improve the quality of healthcare and get earlier recovery and better outcome for patients undergoing THA and TKA, so as to slow the growth of the heavy economic burden associated with the increase of the procedures.

Enhanced recovery after surgery (ERAS) is proposed as a series of evidence-based perioperative optimization with multidisciplinary treatment to reduce surgical stress and accelerate postoperative recovery. Under this general guidelines, different ERAS pathways have been reported to decrease morbidity, save costs, promote faster recovery, and achieve the clinical and economic gain in colorectal, thoracic, and orthopedic surgery. Regional anesthesia was recommended for ERAS because it provides reliable analgesia and little disturbance on hemodynamics in previous literatures. But for patients undergoing THA and TKA, epidural or spinal anesthesia is always associated with indwelling urinary catheter even in surgery with short duration and small amount of blood loss, and femoral or sciatic nerve block decreases muscle strength, leading to postponed mobilization. Nowadays, anesthetic agents with rapid onsetting and clearance make ERAS be applied under general anesthesia. For example, desflurane, a volatile anesthetic with a low blood/gas distribution coefficient, has been reported to metabolized quickly with minor dependence on liver and kidney function, and provide rapid awakening from anesthetic state. Based on its characteristics, we hypothesized that ERAS could be achieved by general anesthesia with the use of short-acting anesthetic agents with the combination of short-acting opioids and muscle relaxant.

In this trial, we'll develop ERAS pathway in patients undergoing primary THA and TKA, and compare with the conventional treatment in length of stay (LOS) in hospital, postoperative complications, as well as the hospitalization costs. The aim of this trial is to verify our hypothesis that ERAS could provide reduced LOS while not increase complications and in-hospital cost when compared with the current clinical practice.

ELIGIBILITY:
Inclusion criteria

* Patients undergoing primary TKA and THA, with both genders.
* Aged more than 18 years.
* Ability to communicate. Exclusion criteria
* Refuse to sign consent.
* Pregnancy or lactating woman
* History or family history of malignant hyperthermia.
* Known allergy to desflurane or any other anesthetic agent.
* History of substance abuse.
* History of postoperative delirium.
* Impairment of cognitive function or communication.
* Psychopathy.
* Active participation in another trial where the primary endpoint follow-up is ongoing.
* Unwillingness or inability to comply with protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay (LOS) in hospital | 30 days
  Time from the day on arrival at hospital to discharge from the hospital (unit: days).

SECONDARY OUTCOMES:
Postoperative LOS | 30 days
  Time from the day of operation to discharge from the hospital (unit: days).
All-cause mortality by 30 days after operation. | 30 days after operation
  All-cause mortality by 30 days after operation.
In-hospital complications | 30 days after operation
  Complications after operation
Mobilization time | 30 days after operation
  Time from the end of operation to ability to walk without human assistance (unit: hours).
Numerical rating scales (NRS) scores at rest and with mobilization or physical therapy | 14 days after operation
  NRS scores will be applied to evaluate the postoperative pain by the patients themselves using a single 11-point numeric rating scale, which is ranged from 0 to 10, where 0 indicates "no pain" and 10 represents "worst imaginable pain".
Postoperative analgesics requirement. | 7 days after operation
  Postoperative sufentanil or other analgesics requirement.
Total in-hospital cost. | 30 days
  All cost during hospitalization
Readmission rate | 30 days after discharge
  Readmission rate by 30 days after discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Principal Investigator — Department of anesthesiology, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be accessed under request to Dr. Ren Liao by email: liaoren7733@163.com.
Supporting Information: Study Protocol
Time Frame: From January 1, 2023 for 5 years.
Access Criteria: Data will be accessed under request to Dr. Ren Liao by email: liaoren7733@163.com.

REFERENCES:
- [Derived] Liao C, Lai X, Zhong J, Zeng W, Zhang J, Deng W, Shu J, Zhong H, Cai L, Liao R. Reducing the length of hospital stay for patients undergoing primary total knee arthroplasty by application of enhanced recovery after surgery (ERAS) pathway: a multicenter, prospective, randomized controlled trial. Eur J Med Res. 2025 May 14;30(1):385. doi: 10.1186/s40001-025-02647-8. PMID 40369602
- [Derived] Li J, Zhu H, Liao R. Enhanced recovery after surgery (ERAS) pathway for primary hip and knee arthroplasty: study protocol for a randomized controlled trial. Trials. 2019 Oct 22;20(1):599. doi: 10.1186/s13063-019-3706-8. PMID 31640757